CLINICAL TRIAL: NCT06934356
Title: Shared Subcortical Arousal Systems Across Perceptual Modalities
Brief Title: Subcortical Arousal in Perceptual Awareness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000037710; 1R01NS134655-01A1 (NIH)
Record Dates: First submitted 2025-03-19; First posted 2025-04-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Electroencephalography; Eye-Tracking Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Thalamic Recording (Aim 1) (Experimental): Participants will perform the visual behavioral task with intracranial electroencephalogram (EEG) brain recordings carried out in parallel with surface EEG recordings. For Aim 1, we will analyze thalamic event related potentials in perceived vs not perceived stimuli, classified as in perception of no report visual stimuli based on eye metrics.
  Interventions: Device: EEG; Device: Eye Tracking; Device: Behavioral task
- Thalamic Stimulation (Aim 2) (Experimental): We will test participants during the Visual Report Paradigm, while recording from the intralaminar thalamus with simultaneous scalp EEG as in Aim 1. Three thalamic stimulation conditions will be tested, randomized across trials: 1. No stimulation; 2. Stimulation Concurrent with visual stimuli; 3. Stimulation Delayed to 2s after visual stimuli. Stimulation will be a 100Hz train lasting 300ms, with biphasic square wave pulses 120μs per phase, current adjusted previously by clinicians to maximum tolerated level without side effects (typically ~3mA).
  The electrical stimulation is being delivered for research purposes to understand the causal role of thalamus in regulating visual perception.
  Interventions: Device: EEG; Device: Eye Tracking; Device: Behavioral task

INTERVENTIONS:
Device: EEG — Participants will have scalp EEG recorded with the international 10-20 system sampled at 256Hz using EEG amplifiers for purposes of surface event related potential analysis
Device: Eye Tracking — An eye-tracking device may be used during the perceptual awareness task. Pupillary and gaze location measurements are recorded using either a ViewPoint~VoltagePro.EyeLink 1000 Plus system, or Argus Science ETVision system. If using the ViewPoint~VoltagePro system or the Argus Science ETVision system, participants will be asked to wear an eye tracker during the perceptual awareness task (similar to wearing sunglasses). If using the EyeLink 1000 Plus system, participants may be asked to place their head inside of a padded head-chin rest to stabilize head position
Device: Behavioral task — For the visual perceptual awareness task, the participant will be presented with barely perceptible visual stimuli. After a variable delay, the participant will be asked to report perception of each stimulus and identify its location.

SUMMARY:
The study is a multi-site study and will be conducted at up to 11 investigative sites in the United States. The study will investigate subcortical arousal circuits in visual perception using techniques with complementary strengths based on promising initial studies.

DETAILED DESCRIPTION:
The study will investigate subcortical arousal circuits in visual perception using techniques with complementary strengths based on promising initial studies. This study is expected to shed important light on the precise relationship between transient increases in subcortical arousal and perceptual awareness, generalizable across the visual modality. This research will therefore provide important general potential benefits, including 1. Identification of subcortical arousal systems in perception, which can benefit treatment of many disorders where perceptual deficits are common, e.g. traumatic brain injury, Alzheimer's disease, stroke, developmental disorders, schizophrenia, epilepsy and others. 2. Understanding the role of specific subcortical arousal circuits in perception may help target improved treatments, including transient thalamic stimulation like that planned for the present investigations, or less invasive treatments (TMS, tDCS, designer drugs) to improve function of these circuits. 3. The planned no-report paradigms may detect perceptual awareness in severe brain damage and anesthesia, where people are unable to overtly respond.

The main hypotheses are that 1. the thalamic awareness potential (TAP) will be associated with visual perception independent of report, and 2. thalamic intralaminar stimulation at the time of stimulus presentation will augment the probability of perceptual awareness.

ELIGIBILITY:
The following are the inclusion/exclusion criteria for epilepsy patients with thalamic electrodes age 13 years and up (Aim 1):

Inclusion Criteria:

* normal vision with or without the use of corrective lenses

Exclusion Criteria:

* severe vision impairment even with correction preventing ability to see stimuli (prevents accurate pupil and eye gaze measurements)
* unable to perform the perception task due to cognitive impairment. All participants must be capable of consenting for themselves.

The following are the inclusion/exclusion criteria for epilepsy patients with thalamic electrodes age 18 years and up (Aim 2):

Inclusion Criteria:

* normal vision with or without the use of corrective lenses
* a female subject must have a negative pregnancy test and if sexually active, must be using a reliable form of birth control for the duration of the trial, be surgically sterile, or be at least two years post-menopausal.

Exclusion Criteria:

* severe vision impairment even with correction preventing ability to see stimuli (prevents accurate pupil and eye gaze measurements)
* unable to perform the perception task due to cognitive impairment. All participants must be capable of consenting for themselves.
* pregnancy

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Subcortical event-related signals | Immediately after the intervention
  Subcortical event-related signals will be recorded by icEEG to assess electrical activity from the cerebral cortex using currently implanted electrodes during the behavioral task
Perceptual Sensitivity | Immediately after the intervention
  measured by the percentage of correctly perceived trials for each participant (Aim 2)

SECONDARY OUTCOMES:
Cortical Event Related Potentials | Immediately after the intervention
  Cortical event related potentials will be measured by scalp EEG to assess brain wave changes at the surface level during the perceptual awareness task

CONTACTS AND LOCATIONS:
Overall Officials: Hal Blumenfeld, MD, Phd, Principal Investigator — Yale University
Locations (8):
- United States (8):
  - Yale School of Medicine, New Haven, Connecticut
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No